CLINICAL TRIAL: NCT00677209
Title: Frankfurt Investigator-initiated Autovaccine-study
Brief Title: The Effect of Autologous Autovaccine in Patients With Allergy on House-dust-mite
Acronym: FIAVS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Prof Stefan Zielen, Childrens Hospital Goethe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVH-2004/1; Eudra-CT Nr. 2005-005534-12
Record Dates: First submitted 2008-05-12; First posted 2008-05-14 (Estimated); Last update posted 2010-12-29 (Estimated); Status verified 2008-05

CONDITIONS: Allergens, House Dust Mites
Keywords: house dust mite; asthma; autovaccine; allergy
MeSH Terms: conditions — Asthma; Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Active Comparator): house dust mite allergics will undergo autovaccine immunization
  Interventions: Biological: Injection of autovaccine (Autovaccine Symbiopharm)

INTERVENTIONS:
Biological: Injection of autovaccine (Autovaccine Symbiopharm) — increasing dosage schedule, six different concentrations, application over six weeks, 2 weeks break, another six weeks, 2 weeks break, than challenge with inhalative house dust mite extract
  Other Names: Autovaccine Symbiopharm

SUMMARY:
House dust mite allergy is a common problem, resulting in asthma, chronic swelling of the eyes, and running nose. The investigators test a possibility to immunize subjects sensitized against house dust mite with extracts from their own gut bacteria "auto-vaccination".

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* age 18-35 years
* known allergy on house-dust mite
* GINA 0-1

Exclusion Criteria:

* anamnestic incompatibility to parts of autovaccine
* asthma > GINA I°
* chronic disease conditions or infections
* pregnancy
* inhalative or systemic steroid use
* any immunosuppressive therapy
* intake of any other probiotic medication (e.g. E.coli nissle 1917)
* participation in any other study at the same time
* substance abuse
* Incapability of understanding the study's purpose and performance
* smoker

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2006-07; Primary Completion 2008-08 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Patients' clinical parameters and behaviour, laboratory values | jul 2006 - august 2008
laboratory testing reflecting function of bone marrow, liver, kidney | jul 2006- august 2008

SECONDARY OUTCOMES:
Lung function,exhalative NO | jul 2006 - oct 2007

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Zielen, M.D., Ph.D., Principal Investigator — Goethe University, Department of pulmonology
Locations (1):
- Goethe University, Department of Pulmonology, Frankfurt am Main, Hesse, Germany

REFERENCES:
- [Background] Halasa J. [Justification of treatment with autovaccine]. Med Dosw Mikrobiol. 1994;46(1-2 Suppl):5-9. No abstract available. Polish. PMID 7967946
- [Derived] Schulze J, Voss S, Zissler U, Rose MA, Zielen S, Schubert R. Airway responses and inflammation in subjects with asthma after four days of repeated high-single-dose allergen challenge. Respir Res. 2012 Sep 19;13(1):78. doi: 10.1186/1465-9921-13-78. PMID 22989372
- [Derived] Rose MA, Weigand B, Schubert R, Schulze J, Zielen S. Safety, tolerability, and impact on allergic inflammation of autologous E.coli autovaccine in the treatment of house dust mite asthma--a prospective open clinical trial. BMC Complement Altern Med. 2011 Jun 3;11:45. doi: 10.1186/1472-6882-11-45. PMID 21639872